CLINICAL TRIAL: NCT04832542
Title: Safety and Effectiveness of Implantable Loop Recorder in Patients With Recurrent, Unexplained, Traumatic Syncope
Brief Title: Implantable Loop Recorder in Traumatic Syncope
Acronym: TRAUMA
Status: Completed | Type: Observational
Sponsor: Azienda Ospedaliera Cardinale G. Panico (Other)
Collaborators: Università Politecnica delle Marche (Other); University of Campania Luigi Vanvitelli (Other); Azienda Ospedaliera Pugliese Ciaccio (Other); Azienda Ospedaliero Universitaria Maggiore della Carita (Other); Cardiology Department, Policlinico Riuniti University Hospital, Foggia, Italy (Unknown); Cardiology Division, Villa Scassi Hospital, Genova ASL 3, Genova (Unknown); San Giuseppe e Melorio Hospital, Santa Maria Capua Vetere (Unknown); Nostra Signora di Bonaria Hospital, San Gavino Monreale (Unknown); Istituto Nazionale di Ricovero e Cura per Anziani (Other)
Responsible Party: Principal Investigator, Pietro Palmisano, MD, Azienda Ospedaliera Cardinale G. Panico
Other Study IDs: TRAUMA
Record Dates: First submitted 2021-04-01; First posted 2021-04-06 (Actual); Last update posted 2021-04-06 (Actual); Status verified 2021-04

CONDITIONS: Syncope
MeSH Terms: conditions — Syncope

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 24 Months
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: outpatient follow-up — The patients were evaluated every six months in order to assess the incidence of traumatic syncope recurrence during follow-up after implantable loop recorder implantation.

SUMMARY:
Prospective, observational registry enrolling consecutive patients with recurrent, unexplained, traumatic syncope underwent implantable loop recorder implantation with the aim to evaluate the incidence of recurrence of traumatic syncope during follow-up.

DETAILED DESCRIPTION:
This observational, prospective registry enrolled consecutive patients with recurrent, unexplained, traumatic syncope underwent implantable loop recorder implantation according to current clinical practice. The patients were evaluated every 6 months based on current clinical practice and the risk of recurrence of traumatic syncope was assessed during follow-up.

ELIGIBILITY:
Inclusion Criteria:

* patients with recurrent, unexplained, traumatic syncope
* patients underwent implantable loop recorder implantation

Exclusion Criteria:

* patients unable to attend scheduled outpatient visits

Min Age: 18 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: Consecutive patients with recurrent, unexplained, traumatic syncope underwent implantable loop recorder implantation
Sampling Method: Probability Sample
Enrollment: 488 (Actual)
Dates: Start 2011-01-01 (Actual); Primary Completion 2020-12-31 (Actual); Study Completion 2021-01-31 (Actual)

PRIMARY OUTCOMES:
Traumatic syncope recurrence | through study completion, an average of 2 year
  Incidence of traumatic syncope recurrence

IPD SHARING:
Plan to Share IPD: No